CLINICAL TRIAL: NCT05323500
Title: Effects of Senobi Breathing Exercises on Body Fat, Lung Functions and Depression in Obese Women
Brief Title: Effects of Senobi Breathing Exercises in Obese Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REC/01292 Sabahat Ali Sheikh
Record Dates: First submitted 2022-04-04; First posted 2022-04-12 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: Quasi experimental Design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Senobi breathing group (Experimental): The study participants will be screened first, then trained to perform SBE (1-minute maneuver). The participants will also guided to repeat this procedure 3 times in one minute with resting period of 10 seconds. They will perform it 3 times a day for 3 months. Assessments will be taken at Baseline & after 3 months.
  Interventions: Other: Senobi breathing exercises

INTERVENTIONS:
Other: Senobi breathing exercises — The study participants will be screened first, then trained to perform SBE (1-minute maneuver). Participants will be instructed to stand upright and tighten their gluteal muscle and then ask them to put one foot in front of their body and placing most of their body weight on back foot. Then, ask them to breath in for three seconds simultaneously, by raising their hands in the air above their heads. After this, instruct them to exhale by using their whole body for pushing air out of the lungs. Participants will also guided to tighten all their body muscles while pushing air out. Exhale should last for seven seconds.

SUMMARY:
Previous studies have been done just in studying the relationship between breathing technique and obesity and described how it proved helpful in decreasing body fat. This study will be very helpful for future researchers as well as in filling the literature gap by explaining the importance of SBE (Senobi Breathing Exercise) in correlation with increased body fat, compromised lung function and depression in females of age from 30 to 60 years.

DETAILED DESCRIPTION:
The study is quasi-experimental study, which is being conducted in a private clinical settings in Khushab. Sample size of 20 individuals was calculated using Hamilton Depression Scale with effect size 0.97 G Power 3.1.9.2 software. The study participants will be screened first, then trained to perform SBE(1-minute maneuver). Participants will be instructed to stand upright and tighten their gluteal muscle and then ask them to put one foot in front of their body and placing most of their body weight on back foot. Then, ask them to breath in for three seconds simultaneously, by raising their hands in the air above their heads. After this, instruct them to exhale by using their whole body for pushing air out of the lungs. Participants will also guided to tighten all their body muscles while pushing air out. Exhale should last for seven seconds. The participants will also guided to repeat this procedure 3 times in one minute with resting period of 10 seconds. They will perform it 3 times a day for 3 months. Assessments will be taken at Baseline & after 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Women of age between 30 to 60 years.
* Asian BMI (> 27.5)
* Obese women with mild to moderate depression

Exclusion Criteria:

* Sedentary lifestyle
* Following an Unhealthy Diet plan
* Any Cardiopulmonary conditions
* Endocrine conditions: hypothyroidism

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Lung volume | changes from Baseline to 3 Months
  Digital spirometry will be used to assess Lung Volumes and capacities
Body Fat | changes from Baseline to 3 Months
  Body Fat Analyzer will be used to assess percent of body fat
waist to hip ratio | changes from Baseline to 3 Months
  Participant is asked to Stand up straight and breathe out. tape measure will be used to check the distance around the smallest part of your waist, just above your belly button. This is waist circumference. Then we will measure the distance around the largest part of your hips - the widest part of your buttocks. This is hip circumference.Waist Hip ratio will be calculated by dividing waist circumference to hip circumference

SECONDARY OUTCOMES:
Hamilton Depression rating Scale | changes from Baseline to 3 Months
  Scoring is based on the 17-item scale and scores of 0-7 are considered as being normal, 8-16 suggest mild depression, 17-23 moderate depression and scores over 24 are indicative of severe depression, the maximum score being 52 on the 17-point scale.

CONTACTS AND LOCATIONS:
Overall Officials: Huma Riaz, PHD*, Principal Investigator — Riphah International University
Locations (2):
- Pakistan (2):
  - Physical Therapy Private Clinic, Khushāb, Punjab Province
  - Pakistan sports complex, Lahore, Punjab Province

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dixon AE, Peters U. The effect of obesity on lung function. Expert Rev Respir Med. 2018 Sep;12(9):755-767. doi: 10.1080/17476348.2018.1506331. Epub 2018 Aug 14. PMID 30056777
- [Background] Mafort TT, Rufino R, Costa CH, Lopes AJ. Obesity: systemic and pulmonary complications, biochemical abnormalities, and impairment of lung function. Multidiscip Respir Med. 2016 Jul 12;11:28. doi: 10.1186/s40248-016-0066-z. eCollection 2016. PMID 27408717
- [Background] Sato K, Kawamura T, Yamagiwa S. The "Senobi" breathing exercise is recommended as first line treatment for obesity. Biomed Res. 2010 Aug;31(4):259-62. doi: 10.2220/biomedres.31.259. PMID 20834183
- [Background] Sato K, Kawamura T, Yamagiwa S. The "Senobi" breathing exercise ameliorates depression in obese women through up-regulation of sympathetic nerve activity and hormone secretion. Biomed Res. 2011 Apr;32(2):175-80. doi: 10.2220/biomedres.32.175. PMID 21551954
- [Background] Sato K, Kawamura T, Abo T. "Senobi" stretch ameliorates asthma symptoms by restoring autonomic nervous system balance. J Investig Med. 2010 Dec;58(8):968-70. doi: 10.231/JIM.0b013e3181f9167b. PMID 20930645